CLINICAL TRIAL: NCT02337166
Title: Regeneration of Human Intrabony Defects With Recombinant Human Fibroblast Growth Factor 2 in a Hyaluronic Acid Gel Carrier - a Longitudinal, Prospective, Randomized Controlled Clinical Trial
Brief Title: Regeneration of Human Intrabony Defects With rhFGF-2/HA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP-HUAM/CCM 21/03
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Periodontitis
Keywords: alveolar bone loss; periodontal attachment loss
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): open instrumentation of the root surfaces and bone defects via flap modified papilla preservation flap
  Interventions: Procedure: Periodontal flap surgery
- Test (Experimental): open instrumentation of the root surfaces and bone defects via flap modified papilla preservation flap and application of a rhFGF-2/HA in the intrabony defect
  Interventions: Device: a gel containing 4mg/ml rhFGF-2 in sodium hyaluronate

INTERVENTIONS:
Device: a gel containing 4mg/ml rhFGF-2 in sodium hyaluronate — 0.2ml of a gel containing 4mg/ml rhFGF-2 in sodium hyaluronate MW 1.3 x 106
  Arms: Test
Procedure: Periodontal flap surgery
  Arms: Control

SUMMARY:
BACKGROUND: Periodontal disease is an infection that results in progressive loss of dental support, which may lead to tooth loss.. The goal of the present study was to evaluate if recombinant human Fibroblast Growth Factor type 2 (rhFGF-2) applied in periodontal intrabony defects in a hyaluronic acid (HA) carrier would enhance the clinical paramenters of regeneration of the periodontal attachment apparatus and the long-term maintenance of the results obtained. METHODS: Thirty adult patients were evaluated. Initial treatment consisted in plaque control measures executed previously to the experimental phase. Two intra-bony defects in each patient were ramdomly allocated for each of the treatment methods employed. Control group (n=30) were treated by open debridement with the papilla preservation flaps, while the text group (n=30) also received a topical application of rhFGF-2/HA in the intrabony defect. The parameters evaluated were, probing depth (PD), gingival recession (REC), probing attachment level (PAL) and probing bone level (PBL). Clinical measurements obtained at baseline and 1, 5 and 10 years after the surgical procedure were compared.

DETAILED DESCRIPTION:
Study Population and Experimental Design The study was designed as a randomized, prospective, split-mouth, controlled clinical trial. It was conducted in accordance with the guidelines of the World Medical Association Declaration of Helsinki (version VI, 2002), after approval of the study design and consent by the Faculty of Medicine, Ethical Committee of Medical Research, Federal Fluminense University (Approval protocol CEP-HUAM/CCM 21/03). Written informed consent was obtained from all subjects. Systemically healthy patients with moderate to advanced chronic periodontitis referred to the Department of Periodontology, Faculty of Dentistry, Federal Fluminense University for periodontal treatment of advanced periodontitis were recruited for and treated in the study.

Inclusion criteria of the study were: (a) adult subjects with chronic periodontitis presenting (b) radiographic evidence alveolar bone loss at the proximal aspect of the tooth, (c) intrabony defect deeper than 4mm, (d) probing pocket depth >6 mm at the site, (e) unremarkable general health according to medical history and clinical judgment, (f) no medications taken for at least six months and no antibiotics taken for twelve months before the beginning of the study. Subjects who have quit the habit of smoking for at least one year before the beginning of the study were considered as non-smokers and, if the other included criteria were met, were included in the present sample. Exclusion criteria for the study were: (a) subjects with "early onset" or aggressive forms of periodontitis, (b) current smokers, (c) presence of significant systemic diseases (i.e., cancer, AIDS, diabetes), (d) clinical evidence of furcation defects, (e) presence of apical radioleucency and (f) previous lack of cooperation with the maintenance program.

Two defects were selected from each patient, and were randomly assigned, immediately before each surgical appointment, by computer generated random sequence allocation to one of the two treatment modalities employed: (a) Control: open instrumentation of the root surfaces and bone defects via flap modified papilla preservation flap; (b) Test: open instrumentation of the root surfaces and bone defects via flap modified papilla preservation flap and application of a rhFGF-2/HA in the intrabony defect. Treatment allocation was registered in an allocation table sheet that was unavailable to the clinical examiner throughout the study. Both the control and test sites were treated at the same surgical appointment and no information on treatment allocation was provided to the patient. All surgical procedures were performed by a single operator, which became aware of the site allocation only after completed root planning and conditioning, and immediately before the application of the growth factor in the test sites. A strict surgical protocol emphasizing careful hard- and soft-tissue management, root debridement, wound stability and infection control was employed (Santana et al 2009; Miranda et al 2013). Nonsurgical infection control was performed in the context of cause- related periodontal therapy and consisted of oral hygiene instructions, scaling and root planing, tooth polishing and plaque control measures performed six months prior to regenerative surgery. Patients were re-evaluated three and six months after the completion of the non-surgical cause-related periodontal therapy and enrolled following the later evaluation appointment.

Clinical Recordings Clinical parameters were assessed using the cemento-enamel junction (CEJ) or, when applicable, another defined landmark, as a fixed reference point. All measurements were recorded using an UNC #15 periodontal probe (PCP-UNC 15, Hu-Friedy, Chicago, IL, USA) by a blinded, trained and calibrated examiner (CMMS), unaware of the treatment provided at baseline and one year after treatment. Measurements were recorded to the nearest mm. Full mouth plaque score (FMPS) was recorded dichotomously as the percentage of total surfaces (four sites per tooth) (O'Leary et al. 1972). BOP was also assessed dichotomously at the same sites, and a full mouth bleeding score was calculated. Recession (REC) was measured as the distance from the CEJ to the gingival margin (GM). Probing depth (PD) was measured as the distance from the GM to the bottom of the gingival sulcus. PD and REC were used to calculate the vertical clinical attachment level (PAL). Under local anesthesia, transgingival probing was performed and the distance between the CEJ and the bottom of the defect (distance CEJ-BD) was also recorded. Clinical measurements obtained at baseline (immediately before surgery) and at twelve months are reported. After debridement of the surgical site, the bottom of the defect (BD) was defined as the distance between cemento-enamel junction and base of the defect. Bone crest level (BC) was measured as the distance between the cementoenamel junction and crest of the defect and the intra-bony defect depth (INTRA) was measured as the subtraction of BC from BD measurements (BD-BC). Moreover, the depth of the three, two and one-wall sub-components of the bony defect were also measured. The primary and secondary outcome variables of the present study were, respectively, change in PAL and bone gain (change in distance CEJ-BD).

In order to ensure the reproducibility and consistency of pre- and post-intervention measurements, examiner calibration was performed before the beginning of the study. Fourteen sites, in seven patients, with probing depths >6 mm were evaluated by the examiner on two separate occasions, 48h apart.

Flap Design Intracrevicular incisions were made and buccal and lingual mucoperiosteal flaps, including at least one tooth mesial and another distal the tooth being treated, were elevated by blunt dissection. Extreme care was taken to preserve the marginal gingiva and inter-dental tissue to achieve better closure of the treated sites. Thus, the defect-associated inter-dental papilla was accessed with papilla preservation ﬂap techniques (Takey 1985, Cortellini et al. 1995, Cortellini et al. 1999) according to indications. A vertical releasing incision was performed at the mesial aspect of the flap whenever necessary to obtain optimized, tensionless, access to the surgical area.

Root and bone defect debridement The bone defect was meticulously debrided with surgical curettes and ultrasonic instruments with special effort to remove all the inflammatory granulation tissue, but with no intention to perforate the cortical bone walls. Thorough root planing was performed with hand (Hu-Friedy, IL, USA), rotary (Intensiv, Grancia, Switzerland) and ultrasonic instruments (Cavitron, Dentisply, USA), to remove subgingival plaque and calculus until all root surfaces attained a hard glassy surface. During the instrumentation, the ﬂaps were slightly elevated, carefully protected with periosteal elevators, and frequently irrigated with saline.

Root conditioning and rhFGF-2 application After instrumentation, the root surfaces were washed with saline solution to remove any remaining detached fragments from the defect and surgical field. Then, a freshly prepared tetracycline hydrochloride paste in saline was applied with gentle circular movements on the instrumented and dried root surfaces of both test and control groups for three minutes. After that, the defect area was carefully rinsed with saline. Finally, on the experimental sites, 0.2ml of a gel containing 4mg/ml rhFGF-2 in sodium hyaluronate MW 1.3 x 106 was applied on the dried root surfaces and bone defect. The flaps were then repositioned and tension-free primary flap closure was obtained using internal mattress, and single interrupted sutures (5.0 Ethicon Sutures, Johnson & Johnson, NJ, USA or Gore-tex Sutures, W.L Gore, AZ, USA).

Post-Operative Treatment The patients were prescribed systemic antibiotic therapy consisting of 200mg of doxycycline***** the day before surgery, followed by 100 mg daily continued until the 20th day after surgery. No surgical dressing was used. The patients were instructed to continue their regular home hygiene care, except in the operated area, which was cleaned by means of gentle topical applications of 0.2% chlorhexidine gluconate (Perioxidin®, Lacer, Barcelona, Spain) in saturated cotton swabs. Patients were instructed not to brush or ﬂoss the surgical area for 4 weeks, when mechanical plaque control was re-instituted. The sutures were removed two weeks after surgery. Hyper-mobile teeth were splinted either before or immediately after the surgical procedure.

Maintenance Schedule Patients were enrolled in a stringent post-operative supportive care programme following surgery (Santana et al 2009). All patients were seen weekly during the first three months and bi-weekly for the next three months. Thereafter, the patients were seen once monthly for the last six-month period of the study. After 1 year, the patients were recalled and re-instructed on proper oral hygiene. Sites were rescaled when indicated.

Radiographic assessments Radiographs were taken with a parallel, standardized, technique at baseline (Eickholz et al. 2004). Radiographs were digitized and analysed using NIH Image Analysis software. The anatomical landmarks for the study included cementum-enamel junction (CEJ), alveolar crest (AC) and base of the defect (BD) (Schei et al. 1959). Radiographic defect depth was measured along the root surface, parallel to the root axis, as the distance between CEJ and BD.

Statistical Analyses Quantitative data were recorded as mean and standard deviations. No data points were missing. Sample size was determined by Power analysis, assuming a standard deviation of the difference of 0.5, which indicated that with a sample of 20 subjects, the study would have >90% power to detect a 1-mm difference in the primary outcome measures PAL gain and CEJ-BD reduction between the two groups. In order to verify the normality of the data, the kurtosis and skewness curves were used. Because all data were considered to be normal for the parameters analysed, Student's paired t-test was used for intra-group (baseline versus 12 months) and inter-group (test versus control) comparisons. The level of significance set at 5% was used in all statistical comparisons performed in the software ProStat (Poly Software International, Pearl River, NY, USA) .

ELIGIBILITY:
Inclusion Criteria:

(a) adult subjects with chronic periodontitis presenting (b) radiographic evidence alveolar bone loss at the proximal aspect of the tooth, (c) intrabony defect deeper than 4mm, (d) probing pocket depth >6 mm at the site, (e) unremarkable general health according to medical history and clinical judgment, (f) no medications taken for at least six months and no antibiotics taken for twelve months before the beginning of the study.

Exclusion Criteria:

(a) subjects with "early onset" or aggressive forms of periodontitis, (b) current smokers, (c) presence of significant systemic diseases (i.e., cancer, AIDS, diabetes), (d) clinical evidence of furcation defects, (e) presence of apical radioleucency and (f) previous lack of cooperation with the maintenance program.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Probing attachment level gain | up to 10 years
Bone level gain | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldo B Santana, DDS,MScD,DSc, Principal Investigator — Federal Fluminense University